CLINICAL TRIAL: NCT00002204
Title: A Phase I, Observer-Blind, Placebo-Controlled Study of the Chiron Vaccine HIV p24/MF59 Administered to Healthy HIV-Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Prevention
Other Study IDs: 095; V24P1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Reference Values; Placebos; AIDS Vaccines; HIV Core Protein p24; HIV Seronegativity; MF59 oil emulsion
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV p24/MF59 Vaccine

SUMMARY:
To evaluate the safety and tolerability of the Chiron vaccine human immunodeficiency virus (HIV) p24(25 or 50 micrograms)/MF59 in healthy HIV-1 seronegative adults. To evaluate the immunogenicity of the HIV p24(50 micrograms)/MF59 vaccine.

DETAILED DESCRIPTION:
This study evaluates the safety and immunogenicity of the Chiron vaccine HIV p24/MF59. In Part A, 15 volunteers are randomly assigned to receive either HIV p24/MF59 or a placebo at 0, 1, and 6 months. 10 volunteers receive the vaccine and 5 volunteers receive the placebo. If no serious adverse events are observed within 1 week after the first injection in these first 15 patients, Part B is initiated. In Part B, 25 volunteers are randomly assigned to receive HIV p24/MF59 or a placebo at 0, 1, and 6 months. 20 volunteers receive the vaccine and 5 volunteers receive the placebo.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Good health as determined by medical history, physical examination, and clinical judgment.
* Negative serology for HIV infection as determined by licensed HIV ELISA test performed within 6 weeks prior to first immunization.
* In vitro Epstein-Barr virus-immortalized cell line from peripheral blood can be established (required for selected Part B volunteers only).

Exclusion Criteria

Co-existing Condition:

Volunteers with the following symptoms or conditions are excluded:

* Significant acute systemic infection.
* Occupational or other responsibilities that would prevent completion of participation in the study.
* Any condition that might interfere with the evaluation of the study objectives.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, autoimmune disease, or any serious chronic illness.
* Evidence of psychiatric or medical history or substance abuse that would adversely affect the volunteer's ability to participate in the trial.
* History of anaphylaxis or other serious adverse reactions to vaccines or vaccine components.

  1. Immunosuppressive medications.
* Live, attenuated vaccine within 60 days of study entry.

NOTE:

* Medically indicated subunit or killed vaccines (e.g., influenza or pneumococcal) are not exclusionary but should be given at least 4 weeks before or after HIV immunizations to avoid potential confusion of adverse reactions.
* Experimental agents within 30 days of study entry.
* HIV vaccine or MF59 adjuvant. Blood products or immunoglobulins in the past 3 months.

Engaging in high-risk behavior within 6 months of study entry, i.e.:

* injection drug use, sexual intercourse without a condom with 4 or more partners or with known iv drug user or HIV+ partner, or newly acquired sexually-transmitted disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton Univ Med Ctr / Ped Infect Disease Div, Omaha, Nebraska, United States